CLINICAL TRIAL: NCT06583941
Title: The Dose-Response Effects of Indena's Virtiva® Plus Ginkgo Biloba Extract on Stress, and Cognitive Performance in Participants Experiencing Heightened Stress
Brief Title: Effects of Indena's Virtiva® Plus Ginkgo Biloba Extract on Stress, and Cognitive Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Applied Science & Performance Institute (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IND072924
Record Dates: First submitted 2024-08-31; First posted 2024-09-04 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Stress; Mood; Cognitive Change
Keywords: Ginkgo Biloba Extract

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low Dose Virtiva Plus (Experimental): One dose (1 capsule) of Virtiva Plus will be consumed twice daily for up to 5 weeks. A single dose contains: 120mg Ginkgo biloba extract (leaf), a minimum of 14.4mg phosphatidylserine, and a minimum of 6mg ginkgo flavonglycosides.
  Interventions: Dietary Supplement: Low Dose Virtiva Plus
- High Dose Virtiva Plus (Experimental): One dose (1 capsule) of Virtiva Plus will be consumed twice daily for up to 5 weeks. A single dose contains: 240mg Ginkgo biloba extract (leaf), a minimum of 28.8mg phosphatidylserine, and a minimum of 12mg ginkgo flavonglycosides.
  Interventions: Dietary Supplement: High Dose Virtiva Plus

INTERVENTIONS:
Dietary Supplement: Low Dose Virtiva Plus — Participants will consume a low dose of Virtiva Plus (120mg) twice daily, for 5 weeks. Prior to receiving their first study treatment, participants will undergo baseline assessments on all study variables. Including computerized cognitive assessment and survey questionnaires. After 4 weeks of supplementation, participants will take one serving of their treatment (120mg of Virtiva Plus) with a normal meal. Three hours later, participants will complete cognitive tests. On a separate day, the same procedure will be repeated, and subjects will take the survey tests.
  Arms: Low Dose Virtiva Plus
Dietary Supplement: High Dose Virtiva Plus — Participants will consume a high dose of Virtiva Plus (240mg) twice daily, for 5 weeks. Prior to receiving their first study treatment, participants will undergo baseline assessments on all study variables. Including computerized cognitive assessment and survey questionnaires. After 4 weeks of supplementation, participants will take one serving of their treatment (240mg of Virtiva Plus) with a normal meal. Three hours later, participants will complete cognitive tests. On a separate day, the same procedure will be repeated, and subjects will take the survey tests.
  Arms: High Dose Virtiva Plus

SUMMARY:
This is a randomized, double-blind, 5-week intervention clinical study that aims to investigate the dose-dependent effects of Virtiva® Plus on stress, and cognitive performance in participants experiencing heightened stress. The occurrence of adverse events in response to daily supplementation of Virtiva® Plus will also be measured. The desired sample size for this study is 24 subjects. To account for potential dropouts, we aim to enroll up to 20% over the desired sample size. Therefore, this study will enroll up to 29 subjects. Subjects will be randomly divided into two study groups: low dose (240 mg/day) or high dose (480 mg/day) of Virtiva® Plus. For both groups, the dose will be divided into two equal servings. Blocked randomization will be deployed in which subjects are divided into blocks of 2 subjects and each subject within a block is randomly assigned to one of the two study groups. Participants will be asked to stop taking alternative supplements used for cognitive enhancement 7 days prior to study related cognitive testing assessments.

DETAILED DESCRIPTION:
Enrollment (Week -4 to Week -3): After obtaining written informed consent participants will undergo screening to ensure they are free of cardiovascular-, neurological-, hepatic-, renal-, metabolic diseases, which will be determined by health history questionnaire. Additionally, as part of screening, participants will be required to have a total Perceived Stress Scale (PSS) score >13 and <27 for moderate stress. If they pass the screening tests, they will be given a battery of cognitive assessment tests as part of a familiarization/acquisition phase of testing on a separate day.

Familiarization/acquisition phase with computerized cognitive testing, (Week -2): Subjects will undergo an abbreviated version (~15 minutes) of the computerized cognitive testing to familiarize with the online platform, testing instructions, and cadence of the tests. After completion of the familiarization procedures, subjects will be randomly assigned to one of two study groups (Virtiva® Plus 240 mg/day or Virtiva® Plus 480 mg/day and will be assigned a subject No./ID in the 100 series starting with "101" and continuing in sequential order until enrollment is met.

Baseline Testing (Week -1 [Day -7 to Day -1]): Prior to receiving their first study treatment, participants will undergo baseline assessments on all study variables. Baseline testing will occur within 7 days of being assigned to their study group. On Day -7, participants will consume a normal breakfast (caffeine and stimulant-free), and undertake a cognitive battery of tests (lasting ~30 min) 3-hours post-breakfast (see these tests under Secondary Endpoints). On Day -6, participants will again consume a normal breakfast, and take multiple survey questionnaires 3-hours post-breakfast (see these tests under Primary Endpoints). Between Days -5 to -1, participants will repeat the survey tests in identical manner on two additional days, for a total of three survey tests taken. The average score of the three survey tests will be used for analysis. The tests may be taken on consecutive days.

Study Treatments (Day 1 to Day 35): Participants will be instructed to start their study treatments on Day 1 and continue supplementation for 35+3 days.

Endpoint Cognitive Tests (Week 4 [Days 26 to 28]): Participants will take one serving of their treatment (120 or 240 mg of Virtiva Plus) with a normal meal. Three hours later, participants will complete all cognitive tests described under the Secondary Endpoints section. These cognitive tests will only be taken on one occasion during these three days (Days 26 to 28).

Endpoint Survey Tests (Week 5 [Days 29 to 35]): On three separate occasions between Day 29 to Day 35, participants will consume a normal breakfast (caffeine and stimulant-free), plus one serving of their treatment (120 or 240 mg of Virtiva Plus). Three hours post breakfast, participants will complete all survey questionnaires described in the Primary Endpoints section on three separate occasions. The average score of the three survey tests will be used for analysis. The tests may be taken on consecutive days.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Aged 50 to 70 years (both limits inclusive)
* Body mass index (BMI) value of 18.5-29.99 kg/m2
* Willing and able to give written informed consent
* Able to read, understand, sign and date the informed consent document (English only)
* Able and willing to comply with the schedule visit(s) and study requirements.
* Willing to consume the investigational study product 2 times per day for 5 weeks.
* Willing to maintain a habitual diet and avoid changes during the study period (for example, intermittent fasting, ketogenic diet, Atkins diet, meatless diet, etc.).
* Willing to cease from consuming cognitive enhancement supplements 7 days prior to and after the study commencement, until the end of the study.

Exclusion Criteria:

* Developmental disability or cognitive impairment that would preclude adequate comprehension of the informed consent form and/or ability to follow study subject requirements and/or record the necessary study measurements.
* History of cardiovascular disease (i.e., myocardial infarction, hypertension, hypercholesterolemia, peripheral vascular disease, other)
* History of neurological disorders (Parkinson's, Amyotrophic lateral sclerosis, epilepsy, spinal cord injury resulting in inability to use upper extremities, other)
* History of gastrointestinal disorders that could lead to uncertain absorption of the study supplements, (i.e., inflammatory bowel disease, ulcerative colitis, Crohn's disease, colostomy, or eating disorder)
* History of kidney or liver disease
* History of metabolic disorders (diabetes, metabolic syndrome, other)
* History or current malignancy
* Receiving chemotherapy agents or radiation treatments
* Diagnosis of a terminal illness
* Pregnancy or has breast fed within 3 months prior to enrollment
* Use of prescription medications that impact digestion (i.e., proton pump inhibitor medications, other)
* History or current alcohol or drug abuse
* Has significant concurrent illnesses (controlled or uncontrolled), such as lupus, hepatitis B/C, HIV, serious mental health illness such as dementia or schizophrenia; psychiatric hospitalization in the past two years, or other, which in the opinion of the investigator, such condition might be aggravated as a result of treatment
* The investigator feels that for any reason the subject is not eligible to participate in the study

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-04-04 (Actual); Study Completion 2025-04-04 (Actual)

PRIMARY OUTCOMES:
Generalized Anxiety Disorder-7 (GAD7) | Pre-Event, 5 weeks Post Event
  The Generalized Anxiety Disorder-7 (GAD-7) is a brief, self-administered screening tool designed to identify probable cases of generalized anxiety disorder and assess its severity in both clinical and research settings. The GAD-7 consists of seven items, each reflecting core symptoms of generalized anxiety disorder as outlined in the Diagnostic and Statistical Manual of Mental Disorders. Respondents rate the frequency of these symptoms over the past two weeks on a 4-point Likert scale, ranging from not at all (0) to nearly every day (3). The total score, which ranges from 0 to 21, provides an indication of the severity of anxiety symptoms, with higher scores corresponding to greater symptom severity. The GAD-7 has demonstrated good reliability and validity across diverse populations.
Perceived Stress Scale - 10 (PSS-10) | Pre-Event, 5 weeks Post Event
  The Perceived Stress Scale is a 10-item questionnaire that measures a participant's perceived stress and the degree to which situations in the participant's life are appraised as stressful. The PSS-10 contains a number of direct queries about current levels of experienced stress. Participants responded to questions on a scale ranging from 0 (never) to 4 (very often), with a higher score indicating more perceived stress
Short Form 36 (SF-36) | Pre-Event, 5 weeks Post Event
  The SF-36 is a questionnaire that measures health-related quality of life. Component analyses showed that there are two distinct concepts measured in the questionnaire - a physical component and a mental dimension. The questionnaire is arranged into 8 categories assessing well-being: physical functioning, limitations due to physical health, limitations to emotional problems, energy/fatigue, emotional well-being, social functioning, pain, and general health Question responses range from 1 to 5 or from 1 to 6 and each response is converted to a score from 0 to 100. For all questions, higher scores demonstrated greater well-being.
Satisfaction with Life Scale (SWLS) | Pre-Event, 5 weeks Post Event
  The Satisfaction with Life Scale (SWLS) is a widely used self-report instrument designed to measure an individual's global cognitive judgments of their life satisfaction. Developed by Diener, Emmons, Larsen, and Griffin in 1985, the SWLS consists of five items, each rated on a 7-point Likert scale ranging from "strongly disagree" (1) to "strongly agree" (7). The total score, ranging from 5 to 35, reflects overall life satisfaction, with higher scores indicating greater satisfaction
Positive emotion, Negative Emotion, Engagement, Relationships, Meaning, and Accomplishment (PERMA Profiler) | Pre-Event, 5 weeks Post Event
  The PERMA Profiler is a comprehensive self-report instrument designed to measure well-being across five key dimensions as outlined in Martin Seligman's PERMA model: Positive Emotion, Engagement, Relationships, Meaning, and Accomplishment. The profiler consists of 23 items, with respondents rating their experiences on an 11-point Likert scale, ranging from "never" (0) to "always" (10). The PERMA Profiler also includes items assessing overall well-being, negative emotion, and physical health. This multidimensional approach allows for a nuanced understanding of well-being, capturing both hedonic and eudaimonic aspects
Dysfunctional Attitudes Scale-17 (DAS-17) | Pre-Event, 5 weeks Post Event
  The Dysfunctional Attitudes Scale-17 (DAS-17) is a self-report instrument used to assess cognitive distortions and maladaptive beliefs that are associated with depression and other psychological disorders. This scale consists of 17 items derived from the original 40-item Dysfunctional Attitudes Scale (DAS), which was designed to measure cognitive vulnerability to depression. Respondents rate each item on a 7-point Likert scale, ranging from "totally agree" to "totally disagree." The DAS-17 focuses on two primary dimensions: perfectionism/performance evaluation and dependency/need for approval. Higher scores on the DAS-17 indicate a greater endorsement of dysfunctional attitudes (Power & Dalgleish, 1997).
Everyday Cognition 12 Scale (ECog-12) | Pre-Event, 5 weeks Post Event
  The Everyday Cognition 12 Scale (ECog-12) is a brief, informant-rated assessment tool designed to measure everyday cognitive function in older adults. Derived from the longer Everyday Cognition (ECog) scale, the ECog-12 focuses on evaluating changes in cognitive abilities that occur in everyday life across multiple domains, including memory, language, visuospatial abilities, planning, organization, and divided attention. Informants rate each of the 12 items based on the observed frequency of cognitive difficulties over the past 10 years, using a 4-point Likert scale ranging from "no change" (1) to "a lot more frequently" (4). The ECog-12 is used in both clinical and research settings to detect early cognitive decline and monitor changes over time (Farias et al., 2008).
Abbreviated Profile of Mood States (POMS) | Pre-Event, 5 weeks Post Event
  The abbreviated POMS as used in this study is a 40-item version where participants rate each item on a 5-point Likert scale with anchors ranging between "Not at all" to "Extremely." The scores are ranked on a scale of 0 to 4. For instance, if you said you are "Not at all" Tense that would score a 0; if you were "Extremely" Tense that would rank a 4. Items are combined to form six separate subscales: tension, depression, anger, vigor, fatigue, and confusion. The subscale scores are then combined to form an overall measure of affect that is labeled as total mood disturbance (TMD). A lower score indicates lower mood disturbance, while a higher score indicates increased mood disturbance.

SECONDARY OUTCOMES:
Visual memory | Pre-Event, 5 weeks Post Event
  The visual memory test measures how well a subject can recognize, remember, and retrieve geometric figures or spatial representations.
Verbal Memory | Pre-Event, 5 weeks Post Event
  The verbal memory test measures how well a subject can recognize, remember, and retrieve words.
Finger Tapping Test (FTT) | Pre-Event, 5 weeks Post Event
  The FTT measures the speed and number of finger-taps on each hand.
Symbol Digit Coding (SDC) | Pre-Event, 5 weeks Post Event
  Measures the speed of processing while drawing upon several cognitive processes simultaneously (i.e., visual scanning, visual perception, visual memory, and motor functions).
Stroop Test | Pre-Event, 5 weeks Post Event
  Assesses the ability to inhibit cognitive interference that occurs when the processing of a stimulus impedes the simultaneous processing of a second stimulus.
Shifting Attention | Pre-Event, 5 weeks Post Event
  Measures a subject's executive function (i.e., rules, categories, decision making) or their ability to shift from one instruction set to another quickly and accurately.
Continuous Performance Test | Pre-Event, 5 weeks Post Event
  Measures vigilance or sustained attention over time.
4-Part Continuous Performance Test (4PCPT) | Pre-Event, 5 weeks Post Event
  The 4PCPT test is a four-part test that measures a participant's working memory and sustained attention.

CONTACTS AND LOCATIONS:
Locations (1):
- The Applied Science and Performance Institute, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared